CLINICAL TRIAL: NCT07118137
Title: Translational Neuroscience CAG for Alzheimer's Disease
Brief Title: Memory Deterioration in Alzheimer Disease
Acronym: MemAD
Status: Recruiting | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 490656
Record Dates: First submitted 2025-08-04; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Alzheimer Disease; Neurodegenerative Diseases; Magnetic Resonance Imaging; Memory Impairment
MeSH Terms: conditions — Alzheimer Disease; Neurodegenerative Diseases; Memory Disorders | interventions — Magnetic Resonance Imaging; Electroencephalography; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — * Blood samples
  * Fecal samples
  All samples will be anonymized and safed according to GDPR and ethical guidelines given by regional ethical commitee.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Mild Alzheimer: Patients above 65 diagnosed with Alzheimer's Disease according to appropriate ICD-criterias.
  Interventions: Device: 7T MRI; Device: EEG; Biological: Blood samples; Biological: Stool samples; Diagnostic Test: Neuropsychologic test (MoCA)
- Controls: Age- and gender-matched control group.
  Interventions: Device: 7T MRI; Device: EEG; Biological: Blood samples; Biological: Stool samples; Diagnostic Test: Neuropsychologic test (MoCA)

INTERVENTIONS:
Device: 7T MRI — Resting and activity-based MRI. Dring activity based MRI, the participant will complete tasks testing semantic memory.
  Other Names: Magnetic Resonance imaging
Device: EEG — Resting-state EEG
  Other Names: Electrophysiology
Biological: Blood samples — Blood samples taken for analysis of central blood biomarkers.
Biological: Stool samples — Stool samples collected to identify distinct gut-microbiota compositions between the groups.
  Other Names: Fecal Speciments
Diagnostic Test: Neuropsychologic test (MoCA) — Map cognition with clinically well-established neuropsychology test

SUMMARY:
Semantic AD

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis based on current ICD criteria for AD or MCI .
* >55years.
* Norwegian native speaker
* Lives at home and not in a health institution

Exclusion Criteria:

* Patients with severe cognitive impairment that prevents assessment with the selected modalities (planned cut-off: CDR > 2).
* Presence of brain tumors.
* History of traumatic brain injury.
* History of cranial surgery.
* Contraindications to the selected imaging modalities (e.g., 7T MRI or EEG).
* Diagnosis of other neurodegenerative diseases such as Parkinson's disease or ALS.

  7T MRI contraindications:
* Large tattoos close to the head region, permanent makeup or unremoveable piercings
* Certain models of pacemakers (if pacemaker implantet, MRI physicist at 7T-lab will be conferred)
* Implantet metal in body (clips, stents, prothesis, skrews, plates, teeth etc.)

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the region of Trøndelag, Norway. The study population will include individuals with cognitive symptoms as well as cognitively healthy, age- and sex-matched controls. Recruitment will take place through memory clinics and primary care services. All participants will undergo standardized assessments and data collection as specified in the study protocol.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-10-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Understand which individual differences are observed among patients with Alzheimer's disease (AD). | From enrollment to end of follow-up at 1 year.
  This outcome will characterize individual variability among patients diagnosed with Alzheimer's disease based on clinical symptoms, cognitive assessments, neuroimaging findings (7T MRI), electrophysiological data (EEG), and biological samples (blood and stool). The goal is to identify patterns or subtypes that may reflect distinct disease mechanisms or progression profiles.
Compare changes in the brain, blood, and stool samples between dementia patients and healthy controls. | From project enrollment to end of follow-up at 1 year.
  Assess differences between dementia patients and cognitively healthy controls using multimodal data, including 7T MRI for brain structure, EEG, blood biomarkers, and gut microbiome profiles from stool samples. The aim is to identify biological and neurological markers associated with dementia-related changes.

SECONDARY OUTCOMES:
Understand which individuals with mild cognitive impairment (MCI) go on to develop Alzheimer's disease (AD). | From enrollment to the end of follow-up time at 1 year.
  Identify early clinical, neuroimaging, and biological markers associated with progression from MCI to AD. This research question aims to improve early diagnosis and risk stratification in individuals with MCI.

OTHER OUTCOMES:
Compare brain changes in patients with Alzheimer's disease (AD) to those with other types of dementia. | From project encrollment to end of follow-up at 1 year.
  This outcome will investigate brain changes in patients with Alzheimer's disease compared to those with other dementia types using the different modalities included in the project.

CONTACTS AND LOCATIONS:
Overall Officials: Axel Sandvig Professor, MD PhD, Principal Investigator — Norwegian University of Science and Technology (NTNU)
Locations (1):
- Norwegian University of Sciene and Technology / Norges teknisk-naturvitenskapelige universitet (NTNU), Trondheim, Trønderlag, Norway

IPD SHARING:
Plan to Share IPD: No
All data will be anonymized.